CLINICAL TRIAL: NCT01190254
Title: An 8-week, Placebo-controlled, Double-blind, Randomized, Fixed-dose Efficacy and Safety Trial of Asenapine in Adolescent Subjects With Schizophrenia
Brief Title: Fixed Dose Efficacy and Safety Study of Asenapine for the Treatment of Schizophrenia in Adolescents (P05896)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05896; 2009-017971-10 (EudraCT Number); MK-8274-020 (Other: Merck Research Laboratories); CTRI/2011/07/001909 (Other: CTRI)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia, Paranoid; Schizophrenia, Disorganized; Schizophrenia, Undifferentiated
Keywords: Asenapine; adolescents; schizophrenia; phase IIIb; placebo-controlled
MeSH Terms: conditions — Schizophrenia, Paranoid; Schizophrenia, Disorganized; Schizophrenia; Disorders of Sex Development | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Asenapine 2.5 mg BID (Experimental): Participants receive active asenapine 2.5 mg tablets sublingually BID for 8 weeks.
  Interventions: Drug: asenapine 2.5 mg
- Asenapine 5.0 mg BID (Experimental): Participants receive active asenapine 2.5 mg tablets sublingually BID through Day 3. On Day 4 participants receive asenapine 2.5 mg in the morning and 5.0 mg in the evening. Participants receive active asenapine 5.0 mg tablets sublingually BID for the remainder of the 8-week treatment period.
  Interventions: Drug: asenapine 2.5 mg; Drug: asenapine 5.0 mg
- Placebo (Placebo Comparator): Participants receive placebo asenapine tablets sublingually BID for 8 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: asenapine 2.5 mg — asenapine 2.5 mg tablets for sublingual administration
  Other Names: Saphris®, SCH 900274, Org 5222
  Arms: Asenapine 2.5 mg BID; Asenapine 5.0 mg BID
Drug: asenapine 5.0 mg — asenapine 5.0 mg tablets for sublingual administration
  Other Names: Saphris®, SCH 900274, Org 5222
  Arms: Asenapine 5.0 mg BID
Drug: placebo — asenapine-matched placebo tablets for sublingual administration
  Arms: Placebo

SUMMARY:
This study is designed to evaluate whether asenapine, which is approved by the United States Food and Drug Administration (US FDA) for acute treatment of schizophrenia in adults, is also effective in adolescents with schizophrenia. Participants who qualify for the study will be randomly assigned to receive a fixed dose of asenapine (either 2.5 mg or 5 mg twice daily [BID]) or placebo for 8 weeks. Throughout the study, observations will be made on each participant at various times to assess the efficacy and safety of the study treatment. The primary objective of the trial is to demonstrate significant superiority of at least one asenapine dose to placebo, as measured by the change from baseline of the Positive and Negative Syndrome Scale (PANSS) total score at Day 56.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must have schizophrenia, diagnosed and confirmed by board-eligible or board certified psychiatrists with at least two years of specialization in pediatric/adolescent psychiatric medicine.
* Each participant must be ≥12 years of age and <18 years of age.
* Each participant must have a minimum PANSS total score of 80 at Screening and Baseline.
* Each participant must have a score of at least 4 (moderate) on two or more of the five items in the positive subscale of the PANSS (delusions, conceptual disorganization, hallucinatory behavior, grandiosity, suspiciousness/ persecution) at Screening and Baseline.
* Each participant must have a CGI-S scale score of ≥4 at Screening and Baseline.
* Each participant must taper off all prohibited psychotropic medications (including antipsychotics, antidepressants, and mood stabilizers) prior to Baseline.
* Each participant must agree not to begin formal, structured psychotherapy during the trial.

Exclusion Criteria:

* A participant must not have a diagnosis of schizoaffective disorder; schizophrenia of residual subtype; schizophrenia of catatonic subtype, or schizophrenia with "continuous," "single episode in partial remission," or "single episode in full remission" course specifiers.
* A participant must not have a primary Axis I diagnosis other than schizophrenia and must not have a comorbid Axis I diagnosis that is primarily responsible for current symptoms and functional impairment.
* A participant must not have a known or suspected diagnosis of mental retardation or organic brain disorder.
* A participant must not currently (within the past 6 months) meet the Diagnostic and Statistical Manual of Mental Disorders-IV-Text Revision (DSM-IV-TR^TM) criteria for substance abuse or dependence (excluding nicotine).
* A participant must not have a diagnosis of psychotic disorder or a behavioral disturbance thought to be substance induced or due to substance abuse.
* A participant must not be at imminent risk of self-harm or harm to others, in the investigator's opinion based on clinical interview and responses provided on the Columbia Suicide Severity Rating Scale (C-SSRS).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2010-09-28 (Actual); Primary Completion 2013-03-10 (Actual); Study Completion 2013-04-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Findling RL, Landbloom RP, Mackle M, Pallozzi W, Braat S, Hundt C, Wamboldt MZ, Mathews M. Safety and Efficacy from an 8 Week Double-Blind Trial and a 26 Week Open-Label Extension of Asenapine in Adolescents with Schizophrenia. J Child Adolesc Psychopharmacol. 2015 Jun;25(5):384-96. doi: 10.1089/cap.2015.0027. PMID 26091193

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants receive placebo asenapine tablets sublingually twice daily (BID) for 8 weeks
Period: Overall Study
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Started | 102 | 98 | 106
Treated | 102 | 98 | 106
Completed | 81 | 81 | 84
Not Completed | 21 | 17 | 22
Not completed — Adverse Event | 3 | 6 | 8
Not completed — Lack of Efficacy | 7 | 4 | 5
Not completed — Lost to Follow-up | 4 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 7
Not completed — Protocol Violation | 2 | 0 | 2
Not completed — Did not meet protocol eligibility | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Total
Number analyzed (Participants) | 102 | 98 | 106 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.4) | 15.2 (1.5) | 15.4 (1.5) | 15.3 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 39 | 115
  Male | 62 | 62 | 67 | 191
Positive and Negative Syndrome Scale (PANSS) total score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score (30 items) ranged from 30 to 210 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (Full Analysis Set [FAS]): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 97.5 (10.3) | 97.4 (10.2) | 98.6 (13.4) | 97.9 (11.4)
Clinical Global Impression of Severity (CGI-S) score [Mean (Standard Deviation); unit: score on a scale] — CGI-S is a 7-point scale for assessing the global severity of the participant's illness, with ratings from 1=normal, not ill to 7=very severely ill. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 4.6 (0.6) | 4.6 (0.6) | 4.7 (0.6) | 4.6 (0.6)
PANSS positive subscale score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS positive subscale score (7 PANSS items) ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 25.5 (3.8) | 25.4 (4.2) | 26.2 (4.5) | 25.7 (4.2)
PANSS negative subscale score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS negative subscale score (7 PANSS items) ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 25.0 (4.5) | 24.9 (4.8) | 24.5 (5.4) | 24.8 (4.9)
PANSS positive and negative subscale scores combined [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS positive and negative subscale scores combined (14 PANSS items) ranged from 14 to 98 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 50.5 (5.7) | 50.2 (5.9) | 50.7 (7.3) | 50.5 (6.3)
PANSS general psychopathology subscale score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS general psychopathology subscale score (16 PANSS items) ranged from 16 to 112 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 47.1 (6.4) | 47.2 (6.0) | 47.9 (7.7) | 47.4 (6.8)
PANSS Marder positive symptoms factor score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder positive symptoms factor score (calculated from value of 8 identified PANSS items) ranged from 8 to 56 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 28.4 (4.0) | 28.7 (3.6) | 28.9 (4.3) | 28.7 (4.0)
PANSS Marder negative symptoms factor score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder negative symptoms factor score (calculated from value of 7 identified PANSS items) ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 24.2 (4.8) | 23.9 (5.4) | 23.8 (5.9) | 23.9 (5.4)
PANSS Marder disorganized thoughts factor score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder disorganized thoughts factor score (calculated from value of 7 identified PANSS items) ranged from 7 to 49 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 22.4 (3.7) | 22.3 (3.4) | 22.5 (4.6) | 22.4 (3.9)
PANSS Marder hostility/excitement factor score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder hostility/excitement factor score (calculated from value of 4 identified PANSS items) ranged from 4 to 28 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 12.9 (3.5) | 12.8 (3.6) | 13.1 (4.3) | 12.9 (3.8)
PANSS Marder anxiety/depression factor score [Mean (Standard Deviation); unit: score on a scale] — The PANSS is a 30-item scale for assessing the symptoms of schizophrenia. For each PANSS item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder anxiety/depression factor score (calculated from value of 4 identified PANSS items) ranged from 4 to 28 with a higher score indicating greater severity of symptoms. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 9.6 (3.1) | 9.8 (3.1) | 10.3 (3.1) | 9.9 (3.1)
Children's Global Assessment Scale (CGAS) score - current functioning [Mean (Standard Deviation); unit: score on a scale] — CGAS is a 100-point scale measuring psychological, social, and school functioning in children aged 6-17. Minimum scores ranged from 1-10, representing the need for constant supervision (worse result) to maximum scores of 91-100, representing superior functioning (better result). Summary statistics presented are for efficacy population (FAS) except as noted: N=99 (baseline value not available for 1 FAS participant in this group), 96, 104 and 299 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 43.0 (8.4) | 41.6 (9.1) | 42.9 (8.5) | 42.5 (8.7)
Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) total score [Mean (Standard Deviation); unit: score on a scale] — PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant is asked to rate 15 items reflecting quality of life with respect to the previous week on a scale of 1=very poor to 5=very good. The PQ-LES-Q total score (sum of Items 1-14) for each participant ranged from 14 to 70 with a higher score indicating better quality of life. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 41.6 (10.7) | 41.2 (10.0) | 40.7 (9.5) | 41.1 (10.1)
PQ-LES-Q overall score [Mean (Standard Deviation); unit: score on a scale] — PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant is asked to rate 15 items reflecting quality of life with respect to the previous week on a scale of 1=very poor to 5=very good. The PQ-LES-Q overall score (Item 15, a global assessment of quality of life) ranged from 1 to 5 with a higher score indicating better quality of life. Summary statistics presented are for efficacy population (FAS): N=100, 96, 104 and 300 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID and Total groups, respectively.
  score on a scale | 3.1 (1.0) | 3.1 (0.9) | 3.0 (1.0) | 3.1 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 56
Description: The PANSS is a 30-item clinician-rated instrument for assessing the symptoms of schizophrenia. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). Positive symptoms refer to an excess or distortion of normal mental status (e.g., delusions). Negative symptoms represent a diminution or loss of normal functions (e.g., emotional withdrawal). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was calculated as the sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy Full Analysis Set [FAS]); also, to be included an on-treatment Day 56 value of PANSS Total Score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -17.8 (17.8) [-20.7 to -13.5] | -23.7 (18.6) [-25.5 to -18.2] | -25.5 (16.9) [-26.3 to -19.1]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.070, Mixed Model for Repeated Measures (MMRM) — p-value is adjusted by Hochberg's method for testing two asenapine groups versus the placebo group; Model included terms of (pooled) site, treatment, visit, baseline, and the interaction of visit by treatment and baseline by visit; Difference in Least Squares (LS) Means = -4.8, 95% CI 2-sided [-9.9 to 0.4] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.064, MMRM — p-value is adjusted by Hochberg's method for testing two asenapine groups versus the placebo group; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -5.6, 95% CI 2-sided [-10.7 to -0.5] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID; Investigation of dose-response relationship of change from baseline to Day 56 in PANSS Total Score was a Secondary study endpoint. Multiple contrast testing using MMRM model was used to evaluate 3 pre-defined dose-response patterns (Linear, Convex, Concave); Test type: Superiority or Other; p = 0.064, MMRM — p-value (adjusted to control Type I error in multiple testing) for Linear dose-response pattern (Placebo<2.5 mg<5.0 mg)
Statistical Analysis 4: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.046, MMRM — p-value (adjusted to control Type I error in multiple testing) for Convex dose-response pattern (Placebo<2.5 mg=5.0 mg)
Statistical Analysis 5: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.273, MMRM — p-value (adjusted to control Type I error in multiple testing) for Concave dose-response pattern (Placebo=2.5 mg<5.0 mg)

2. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at Day 56
Description: Change from baseline in CGI-S score at Day 56 is the Key Secondary Outcome Measure. CGI-S is a 7-point scale for assessing the global severity of the participant's illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the CGI-S score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 76 | 72 | 79
score on a scale | -0.8 (1.1) [-1.0 to -0.6] | -1.1 (1.0) [-1.2 to -0.8] | -1.3 (1.0) [-1.4 to -1.0]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Confirmative testing for the key secondary endpoint was to be performed only if both asenapine doses were superior to placebo in change from baseline in PANSS total score at Day 56 (hypotheses associated with Primary outcome measure). If this did not occur, no confirmative testing could be performed and multiplicity unadjusted p-values are provided. Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.218, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.2, 95% CI 2-sided [-0.5 to 0.1] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.024, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.3, 95% CI [-0.6 to -0.0] — Estimate is asenapine versus placebo

3. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score at Day 56
Description: This measure reports results for the 7 items of the positive subscale of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal mental status (e.g., delusions). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS positive subscale score for each participant was calculated as the sum of the rating assigned to each of the 7 subscale items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS positive subscale score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -6.0 (6.1) [-7.1 to -4.7] | -7.9 (5.8) [-8.7 to -6.3] | -9.1 (5.6) [-9.3 to -6.9]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.067, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.6, 95% CI 2-sided [-3.3 to 0.1] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.012, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.1, 95% CI 2-sided [-3.8 to -0.5] — Estimate is asenapine versus placebo

4. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score at Day 56
Description: This measure reports results for the 7 items of the negative subscale of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions (e.g., emotional withdrawal). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS negative subscale score for each participant was calculated as the sum of the rating assigned to each of the 7 subscale items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS negative subscale score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -3.4 (5.2) [-4.3 to -2.3] | -4.8 (5.6) [-5.5 to -3.5] | -4.9 (4.5) [-5.5 to -3.5]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.097, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.2, 95% CI 2-sided [-2.6 to 0.2] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.099, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.2, 95% CI 2-sided [-2.6 to 0.2] — Estimate is asenapine versus placebo

5. Secondary Outcome: Change From Baseline in PANSS Positive and Negative Subscale Scores Combined at Day 56
Description: This measure reports results for the combined positive subscale (7 items) and negative subscale (7 items) of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal mental status (e.g., delusions). Negative symptoms represent a diminution or loss of normal functions (e.g., emotional withdrawal). For each of the total 14 items in the combined positive and negative subscales, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS positive and negative subscale scores combined for each participant was calculated as the sum of the rating assigned to each of the 14 combined subscale items, and ranged from 14 to 98 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS positive/negative subscale scores combined must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -9.4 (10.1) [-11.2 to -7.2] | -12.7 (10.2) [-14.0 to -9.9] | -14.0 (8.8) [-14.4 to -10.5]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.062, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.7, 95% CI 2-sided [-5.6 to 0.1] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.025, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -3.2, 95% CI 2-sided [-6.0 to -0.4] — Estimate is asenapine versus placebo

6. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscale Score at Day 56
Description: This measure reports results for the 16 items of the general psychopathology subscale of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS general psychopathology subscale score for each participant was calculated as the sum of the rating assigned to each of the 16 subscale items, and ranged from 16 to 112 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS general psychopathology subscale score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -8.5 (8.6) [-9.7 to -6.2] | -10.9 (9.5) [-11.9 to -8.3] | -11.5 (8.9) [-12.0 to -8.5]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.098, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.1, 95% CI 2-sided [-4.6 to 0.4] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.071, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.3, 95% CI 2-sided [-4.8 to 0.2] — Estimate is asenapine versus placebo

7. Secondary Outcome: Change From Baseline in PANSS Marder Positive Symptoms Factor Score at Day 56
Description: This measure reports results for the 8 items of the Marder positive symptoms factor of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. Marder factors are a modified grouping of the 30 PANSS items (Marder et al. J Clin Psychiatry 1997;58(12):538-46). Positive symptoms refer to an excess or distortion of normal mental status (e.g., delusions). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder positive symptoms factor score for each participant was calculated as the sum of the rating assigned to each of the 8 applicable Marder factor items, and ranged from 8 to 56 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS Marder positive symptoms factor score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -6.1 (6.1) [-7.3 to -4.9] | -7.9 (6.1) [-8.7 to -6.2] | -8.9 (5.5) [-9.2 to -6.8]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.106, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.4, 95% CI 2-sided [-3.1 to 0.3] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.026, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.9, 95% CI 2-sided [-3.6 to -0.2] — Estimate is asenapine versus placebo

8. Secondary Outcome: Change From Baseline in PANSS Marder Negative Symptoms Factor Score at Day 56
Description: This measure reports results for the 7 items of the Marder negative symptoms factor of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. Marder factors are a modified grouping of the 30 PANSS items. Negative symptoms represent a diminution or loss of normal functions (e.g., emotional withdrawal). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder negative symptoms factor score for each participant was calculated as the sum of the rating assigned to each of the 7 applicable Marder factor items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS Marder negative symptoms factor score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -3.7 (5.3) [-4.6 to -2.6] | -5.2 (5.5) [-5.9 to -3.9] | -5.3 (4.5) [-5.9 to -3.9]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.083, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.2, 95% CI 2-sided [-2.6 to 0.2] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.067, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.3, 95% CI 2-sided [-2.7 to 0.1] — Estimate is asenapine versus placebo

9. Secondary Outcome: Change From Baseline in PANSS Marder Disorganized Thoughts Factor Score at Day 56
Description: This measure reports results for the 7 items of the Marder disorganized thoughts factor of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. Marder factors are a modified grouping of the 30 PANSS items. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder disorganized thoughts factor score for each participant was calculated as the sum of the rating assigned to each of the 7 applicable Marder factor items, and ranged from 7 to 49 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS Marder disorganized thoughts factor score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -3.4 (4.1) [-4.3 to -2.6] | -4.3 (4.3) [-5.2 to -3.5] | -4.8 (4.3) [-5.2 to -3.5]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.131, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.9, 95% CI 2-sided [-2.1 to 0.3] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.135, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.9, 95% CI 2-sided [-2.1 to 0.3] — Estimate is asenapine versus placebo

10. Secondary Outcome: Change From Baseline in PANSS Marder Hostility/Excitement Factor Score at Day 56
Description: This measure reports results for the 4 items of the Marder hostility/excitement factor of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. Marder factors are a modified grouping of the 30 PANSS items. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder hostility/excitement factor score for each participant was calculated as the sum of the rating assigned to each of the 4 applicable Marder factor items, and ranged from 4 to 28 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS Marder hostility/excitement factor score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -2.8 (4.0) [-3.3 to -1.8] | -3.8 (3.6) [-4.3 to -2.8] | -3.8 (4.3) [-4.1 to -2.6]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.071, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.0, 95% CI 2-sided [-2.0 to 0.1] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.120, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.8, 95% CI 2-sided [-1.9 to 0.2] — Estimate is asenapine versus placebo

11. Secondary Outcome: Change From Baseline in PANSS Marder Anxiety/Depression Factor Score at Day 56
Description: This measure reports results for the 4 items of the Marder anxiety/depression factor of the PANSS, which is a 30-item clinician-rated instrument used to assess the symptoms of schizophrenia. Marder factors are a modified grouping of the 30 PANSS items. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS Marder anxiety/depression factor score for each participant was calculated as the sum of the rating assigned to each of the 4 applicable Marder factor items, and ranged from 4 to 28 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at Day 56; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the PANSS Marder anxiety/depression factor score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 77 | 72 | 79
score on a scale | -1.8 (2.4) [-2.3 to -1.2] | -2.4 (2.9) [-2.7 to -1.6] | -2.7 (2.9) [-2.8 to -1.8]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.263, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.4, 95% CI 2-sided [-1.2 to 0.3] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.146, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.5, 95% CI 2-sided [-1.3 to 0.2] — Estimate is asenapine versus placebo

12. Secondary Outcome: Total PANSS 30% Responders
Description: A Total PANSS 30% responder was defined as a participant who had a reduction from baseline of at least 30% in the PANSS Total score at the last available assessment of the study for that participant (i.e., endpoint). The PANSS is a 30-item clinician-rated instrument for assessing the symptoms of schizophrenia. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The Total score is the sum of the ratings for the individual items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms.
Time Frame: Baseline up to Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS).
Measure: Number; unit: participants
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 100 | 96 | 104
participants | 36 | 48 | 51
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.028, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of (pooled) site, treatment, and baseline PANSS Total Score; Odds Ratio (OR) = 2.0, 95% CI 2-sided [1.1 to 3.6] — OR was adjusted for baseline and (pooled) site. An OR of >1 is considered to mean that asenapine has a higher probability of achieving Total PANSS 30% response
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.048, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of (pooled) site, treatment, and baseline PANSS Total Score; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.0 to 3.3] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Kaplan-Meier Estimate of Cumulative Percentage of Participants With Total PANSS 30% Response at End of Study
Description: A total PANSS 30% response was defined as a reduction from baseline of at least 30% in the PANSS Total score. The PANSS is a 30-item clinician-rated instrument for assessing the symptoms of schizophrenia. For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The Total score is the sum of the ratings for the individual items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. The Kaplan-Meier estimate reports the cumulative percentage of participants with total PANSS 30% response from first drug intake up to approximately Day 59.
Time Frame: Baseline up to approximately Day 59
Population: as for outcome 12
Measure: Number; unit: cumulative % of participants w/ Response
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 100 | 96 | 104
cumulative % of participants w/ Response | 62.0 | 64.2 | 72.1
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.576, Log Rank — p-value is for Log Rank test of difference in time to event (PANSS 30% response) curves between the three treatment groups
Statistical Analysis 2: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.171, Regression, Cox; Model included factors for (pooled) site, treatment and baseline PANSS Total Score; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.9 to 2.0] — An HR of >1 is considered to mean that asenapine has a higher likelihood of being a Total PANSS 30% Responder than placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.368, Regression, Cox; Model included factors for (pooled) site, treatment and baseline PANSS Total Score; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.8 to 1.8] — [estimate comment as in outcome 13, analysis 2]

14. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Score at Day 56
Description: CGI-I is a 7-point scale for assessing the global improvement of the participant's illness relative to baseline, with ratings from 1=very much improved to 7=very much worse.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included an on-treatment Day 56 value of the CGI-I score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 76 | 72 | 79
score on a scale | 3.1 (1.1) [2.9 to 3.4] | 2.8 (1.1) [2.7 to 3.1] | 2.5 (1.0) [2.5 to 2.9]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.094, MMRM; Model included terms of (pooled) site, treatment, visit, and the interaction of visit by treatment; Difference in LS Means = -0.3, 95% CI 2-sided [-0.6 to 0.0] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.003, MMRM; Model included terms of (pooled) site, treatment, visit, and the interaction of visit by treatment; Difference in LS Means = -0.5, 95% CI 2-sided [-0.8 to -0.2] — Estimate is asenapine versus placebo

15. Secondary Outcome: CGI-I Responders
Description: A CGI-I responder was defined as a participant who had a CGI-I score of 1 (very much improved) or 2 (much improved) at the last available assessment of the study for that participant (i.e., endpoint). CGI-I is a 7-point scale for assessing the global improvement of the participant's illness relative to baseline, with ratings from 1=very much improved to 7=very much worse.
Time Frame: Baseline up to Day 56
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 100 | 96 | 104
participants | 28 [-7.1 to -4.7] | 36 [-8.7 to -6.3] | 41 [-9.3 to -6.9]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.177, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of region (Asia-Pacific, North America, Eastern Europe [Africa/Latin America sites assigned to this region]) and treatment; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.8 to 2.8] — OR was adjusted for region. An OR of >1 is considered to mean that asenapine has a higher probability of achieving CGI-I response
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.114, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.9 to 2.9] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: Kaplan-Meier Estimate of Cumulative Percentage of Participants With CGI-I Response at End of Study
Description: CGI-I response was defined as the occurrence of a CGI-I score of 1 (very much improved) or 2 (much improved). CGI-I is a 7-point scale for assessing the global improvement of the participant's illness relative to baseline, with ratings from 1=very much improved to 7=very much worse. The Kaplan-Meier estimate reports the cumulative percentage of participants with CGI-I response from first drug intake up to approximately Day 58.
Time Frame: Baseline up to approximately Day 58
Population: as for outcome 12
Measure: Number; unit: cumulative % of participants w/ Response
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 100 | 96 | 104
cumulative % of participants w/ Response | 54.7 | 47.1 | 60.1
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.057, Log Rank — p-value is for Log Rank test of difference in time to event (CGI-I response) curves between the three treatment groups
Statistical Analysis 2: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.135, Regression, Cox; Model included factors for (pooled) site and treatment; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.9 to 2.3] — An HR of >1 is considered to mean that asenapine has a higher likelihood of being a CGI-I Responder than placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.010, Regression, Cox; Model included factors for (pooled) site and treatment; Hazard Ratio (HR) = 1.8, 95% CI 2-sided [1.2 to 2.9] — An HR of >1 is considered to mean that asenapine has a higher likelihood of being a CGI-I Responder than placebo

17. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS) Score at Day 56
Description: CGAS is a 100-point scale measuring psychological, social, and school functioning in children aged 6-17. Minimum scores ranged from 1-10, representing the need for constant supervision (worse result) to maximum scores of 91-100, representing superior functioning (better result). The reported measure is the change from baseline at Day 56; improvement in functioning is represented by positive values.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 56 value of the CGAS score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 76 | 72 | 79
score on a scale | 10.2 (12.9) [7.5 to 12.3] | 12.8 (12.1) [8.9 to 13.7] | 15.0 (10.8) [11.6 to 16.4]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.417, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 1.4, 95% CI 2-sided [-2.0 to 4.8] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Model uses efficacy FAS population (number of participants: placebo - 100, asenapine 2.5 mg - 96, asenapine - 104); Test type: Superiority or Other; p = 0.017, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 4.2, 95% CI 2-sided [0.8 to 7.6] — Estimate is asenapine versus placebo

18. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Total Score at Day 56
Description: PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant is asked to rate 15 items reflecting quality of life with respect to the previous week on a scale of 1=very poor to 5=very good. Items 1-14 assess specific areas (e.g., your health, your mood or feelings); Item 15 is a global assessment of overall quality of life. The PQ-LES-Q total score for each participant was calculated as the sum of the rating assigned to each of the first 14 items, and ranged from 14 to 70 with a higher score indicating better quality of life. The reported measure is the change from baseline at Day 56; improvement in quality of life is represented by positive values. This analysis used a last-observation-carried-forward (LOCF) approach; if no Day 56 value was available for a participant, the last available assessment prior to the Day 56 assessment was used.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and at least 1 post-baseline on-treatment value of the PQ-LES-Q total score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 85 | 83 | 82
score on a scale | 3.1 (8.9) [1.8 to 4.9] | 3.9 (9.3) [2.4 to 5.5] | 6.1 (8.7) [3.9 to 7.0]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.600, ANCOVA; Model included terms of (pooled) site, treatment, and baseline; Difference in LS Means = 0.6, 95% CI 2-sided [-1.6 to 2.8] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.064, ANCOVA; Model included terms of (pooled) site, treatment, and baseline; Difference in LS Means = 2.1, 95% CI 2-sided [-0.1 to 4.3] — Estimate is asenapine versus placebo

19. Secondary Outcome: Change From Baseline in PQ-LES-Q Overall Score (i.e., Item 15) at Day 56
Description: PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant is asked to rate 15 items reflecting quality of life with respect to the previous week on a scale of 1=very poor to 5=very good. Items 1-14 assess specific areas (e.g., your health, your mood or feelings); Item 15 is a global assessment of overall quality of life. The Item 15 result is defined to be the PQ-LES-Q overall score, and ranged from 1 to 5 with a higher score indicating better quality of life. The reported measure is the change from baseline at Day 56; improvement in quality of life is represented by positive values. This analysis used an LOCF approach; if no Day 56 value was available for a participant, the last available assessment prior to the Day 56 assessment was used.
Time Frame: Baseline and Day 56
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment PANSS Total Score (this group is termed the efficacy FAS); also, to be included a baseline and at least 1 post-baseline on-treatment value of the PQ-LES-Q overall score score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Number analyzed (Participants) | 85 | 83 | 82
score on a scale | 0.2 (1.0) [0.1 to 0.4] | 0.3 (1.1) [0.2 to 0.5] | 0.5 (0.9) [0.2 to 0.6]
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.407, ANCOVA; Model included terms of (pooled) site, treatment, and baseline; Difference in LS Means = 0.10, 95% CI 2-sided [-0.13 to 0.33] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.111, ANCOVA; Model included terms of (pooled) site, treatment, and baseline; Difference in LS Means = 0.19, 95% CI 2-sided [-0.04 to 0.42] — Estimate is asenapine versus placebo

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID
Serious Adverse Events (participants affected / at risk) | 3/102 | 3/98 | 3/106
Other Adverse Events (participants affected / at risk) | 23/102 | 39/98 | 46/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | Asenapine 2.5 mg BID (N=98) | Asenapine 5.0 mg BID (N=106)
Schizophrenia (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=102) | Asenapine 2.5 mg BID (N=98) | Asenapine 5.0 mg BID (N=106)
Somnolence (Nervous system disorders) | 7 (7) | 20 (22) | 18 (21)
Headache (Nervous system disorders) | 6 (7) | 7 (12) | 8 (11)
Sedation (Nervous system disorders) | 2 (2) | 4 (4) | 12 (14)
Akathisia (Nervous system disorders) | 1 (1) | 4 (5) | 7 (9)
Dizziness (Nervous system disorders) | 1 (1) | 7 (7) | 2 (5)
Insomnia (Psychiatric disorders) | 6 (8) | 5 (6) | 10 (12)
Nausea (Gastrointestinal disorders) | 8 (9) | 2 (2) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 5 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is planned to first publish/present trial results together with the other sites, unless permission is obtained from Sponsor to publish separate results. Sponsor must be able to review all proposed results communications regarding study 45 days prior to submission for publication/presentation. If there is disagreement concerning appropriateness of the materials, Investigator and Sponsor must meet to make a good faith effort to discuss/resolve disagreement prior to submission for publication.